CLINICAL TRIAL: NCT04732767
Title: Prospective Study of Maternal and Umbilical Cord Blood Collection to Evaluate for Presence of COVID-19 Antibody Response in COVID-19 Positive Women
Brief Title: Evaluation of COVID-19 IgG Antibodies in Maternal and Cord Blood Samples
Status: Withdrawn | Type: Observational
Why Stopped: not enough research personnel to complete study at the time
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 08-20-20E
Record Dates: First submitted 2021-01-28; First posted 2021-02-01 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Pregnancy Related; Antibody Response
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples obtained during the study will include maternal and cord blood samples. These samples will be stored for potential future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Protocol Summary

Study design: Prospective cohort study of pregnant COVID-19 positive patients at delivery.

Study Objective: To collect umbilical cord blood and placenta samples at the time of delivery in COVID-19 positive women and evaluate for presence of COVID-19 virus and maternal antibody response.

Inclusion/Exclusion Criteria: Women admitted for delivery who are known or suspected COVID-19 positive who have had standard nasal swab testing for COVID-19.

Study Procedures: Informed consent for patients will be obtained. Maternal blood will be collected for viral and antibody tests for COVID-19. Following delivery of the neonate, cord blood and placenta samples will be collected and sent for viral PCR and maternal antibody analysis. Neonatal testing will be done as per existing clinical protocol for infants born to PUI/COVID-19 positive women.

Statistical Analysis: Statistical analysis for this study will include descriptive analysis and quantitative statistics of findings.

DETAILED DESCRIPTION:
Background

The clinical syndrome of coronavirus 2019 (COVID-19), caused by the severe acute respiratory 2 virus (SARS-CoV-2) first began in Wuhan China in December 2019 and subsequently spread globally at an exponential rate. The disease was officially classified by the World Health Organization as a pandemic on March 11, 2020. The first death from COVID-19 was reported in the United States on February 28, 2020.

In general, pregnancy is a state of relative immunosuppression, and alterations in immunology and physiology during pregnancy increase the risks of significant respiratory complications and associated obstetrical complications from severe illness. To date, data to guide understanding of the impact of COVID-19 on pregnancy is relatively limited. With any viral illness in pregnancy, there is potential for maternal-fetal transmission. As of now, there have been very few reported cases of suspected vertical transmission. Moreover, there have been few cases of neonatal transmission, even in patients acutely ill with COVID-19 at the time of delivery. However, a recent case report highlighted a 19 week pregnancy loss in a COVID-19 positive patient where placenta pathology showed presence of COVID-19 by PCR, although fetal samples were negative.

As the United States begins to expand testing from viral to antibody testing, opportunity exists to determine if maternal antibodies are present in neonates. If present, these antibodies may confer protection for neonates born to infected mothers. During the course of any infection, IgM antibodies are formed with subsequent development of IgG antibodies. Regardless of source, maternal IgM antibodies do not readily cross the placenta barrier, while maternal IgG antibodies easily cross the placenta during pregnancy. Fetuses are capable of initiating an IgM response to infection in utero. Cord blood serves as a non-invasive source of neonatal blood that can be easily obtained at delivery and allows assessment of the neonate.

Hypothesis

We hypothesize that cord blood collected from COVID-19 positive women will show presence of IgG antibodies against COVID-19 which may confer protection for the infant in the neonatal period.

Objective

To collect: 1. maternal blood samples for COVID-19 IgG antibodies on admission to labor and delivery; 2. cord blood samples for COVID-19 IgG antibodies at the time of delivery; 3. placenta pathology.

Study Type:

Prospective cohort study of pregnant COVID-19 positive patients at delivery admission or at any point during the pregnancy.

Study Methods:

Eligible patients will be invited to participate in the study during pregnancy or on admission to labor and delivery. Eligible patients will have had a positive COVID-19 PCR test at some time during pregnancy or on the delivery admission. Informed consent will be obtained by admitting physician from patients who agree to participate. A maternal blood sample will be obtained with routine admission labs by nursing staff. This sample will be sent for immunoassay for qualitative assessment for COVID-19 IgG antibodies. C-reactive protein will also be measured as this is an indicator of severe disease. At delivery, cord blood and placenta samples will be obtained as per routine collection methods by the delivery physician. Cord blood will be sent for the same analysis as the maternal blood sample. The placenta will be sent to pathology. Results will be obtained through the patient's medical record. Data will be collected into a Redcap database by research personnel. Neonatal data will be obtained from the neonate's medical record and entered into the Redcap database by research personnel. Any publications resulting from this study will use de-identified patient data.

The benefit of this study will be contribution to the limited data that exists around COVID-19 infection and pregnancy.

Data Analysis

Statistical analysis for this study will include descriptive analysis and quantitative statistics of findings.

ELIGIBILITY:
Inclusion Criteria:

- Women admitted for delivery who are known or suspected COVID-19 positive and women were positive at any time during pregnancy who have had standard nasal swab PCR testing for COVID-19.

Exclusion Criteria:

- Patients less than 18 years of age. Patients unable to give consent. Patients who are immunocompromised.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant
Study Population: Pregnant patients at greater than age 18 who have had a positive COVID-19 PCR test during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Presence of COVID-19 IgG antibodies by immunoassay in maternal and cord blood samples. | 6 months
  Immunoassay will be used to detect qualitative levels of COVID-19 IgG antibodies in maternal and cord blood.

CONTACTS AND LOCATIONS:
Overall Officials: Ngina K Connors, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No